CLINICAL TRIAL: NCT00589147
Title: A Prospective, Randomized, Controlled Study Comparing Three Tibial Component Designs in Total Knee Arthoplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Zimmer Biomet (Industry)
Responsible Party: Mark W. Pagnano, MD, Mayo Clinic Rochester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2320-02
Record Dates: First submitted 2007-12-21; First posted 2008-01-09 (Estimated); Last update posted 2012-05-28 (Estimated); Status verified 2012-05

CONDITIONS: Total Knee Arthroplasty

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): One study group will consist of patients treated with the modular cemented tibia.
  Interventions: Device: The Zimmer NexGen Legacy Knee System, modular cemented tibia
- 2 (Active Comparator): Study arm will consist of patients that are treated with non-modular cemented tibia.
  Interventions: Device: The Zimmer NexGen Legacy Knee System, non-modular cemented tibia.
- 3 (Active Comparator): Study arm will consist of patients that are treated with non-modular uncemented tibia.
  Interventions: Device: The Zimmer NexGen Legacy Knee System, non-modular uncemented tibia

INTERVENTIONS:
Device: The Zimmer NexGen Legacy Knee System, modular cemented tibia — modular cemented tibia
  Arms: 1
Device: The Zimmer NexGen Legacy Knee System, non-modular cemented tibia. — non-modular cemented tibia.
  Arms: 2
Device: The Zimmer NexGen Legacy Knee System, non-modular uncemented tibia — non-modular uncemented tibia
  Arms: 3

SUMMARY:
SUMMARY A prospective, randomized, single-blinded clinical trial is proposed to compare three tibial tray designs for patients undergoing total knee arthroplasty. This study is designed to address the clinically important issues of tibial component modularity and fixation in total knee replacement. The Zimmer NexGen Legacy knee system is an FDA approved device and in this study will be used with 1) a modular tibial tray inserted with cement and 2) a non-modular tibial tray inserted with cement, and 3) a non-modular tibial tray inserted without cement. The insertion of total knee components without cement has been done clinically for over 20 years but has not been specifically approved by the FDA. Thus treatment arm 3, a non-modular tray inserted without cement, would involve the so-called off-label use of the device.

136 cases will be assigned to each arm of the study. Each patient will be assessed two months after surgery, one year after surgery, two years after surgery, five years after surgery, and every three to five years thereafter. The principal outcome measures will be the Knee Society Clinical rating scale, the SF-36 and the presence of significant lucent lines.. These measures will be compared among patients in the 3 trial arms at 5 years post surgery (or at the last follow-up point for those who drop out or become lost to follow-up). The Knee Society scores and SF-36 scores will be analyzed using analysis of variance models Rates of significant lucencies, perioperative mortality, as well as complications such as deep vein thrombosis, pulmonary embolus, neurovascular complication, and infection will be compared among the groups using chi-square tests . Rates of revision surgery will be compared among the groups using survivorship methods.

PURPOSE The primary aim of the study is to compare the results obtained with each of three tibial designs for patients undergoing total knee arthroplasty. Those results will be measured with disease-specific (Knee Society Scores), global (SF-36), and outcome measures. Radiographic results consisting of standing alignment, lateral and skyline views of the surgical knee will be recorded and analyzed. Completion of the intial investigation will occur at the 5-year interval after the last enrolled patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients greater then or equal to 20 and less then or equal to 85 undergoing unilateral primary knee surgery for degenerative joint disease (DJD).

Exclusion Criteria:

* Age less than 20 years or > 85.
* Severe deformity great then or equal to 20 degrees varus, valgus malalignment or flexion deformity.
* Osteomyelitis, septicemia, prior infection of knee joint, or other active infections that may spread to other areas of the body.
* The presence of infections, highly communicable diseases, e.g. AIDS, active tuberculosis, venereal disease, and hepatitis.
* Significant neurological or musculoskeletal disorders or disease that may adversely affect normal gait or weight bearing.
* Metastatic disease.
* Any congenital, developmental, or other bone disease or previous knee surgery that may, in the surgeon's judgement, interfere with TK prosthesis survival or success, e.g. Paget's disease, Charcot's disease secondary to diabetes, severe osteoporosis, previous high tibial osteotomy, etc.
* Presence of previous prosthetic knee replacement device (any type).
* Arthrodesis of the affected knee.
* Patients not requiring patella resurfacing.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 397 (Actual)
Dates: Start 2003-08; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
The primary aim of the study is to compare the results obtained with each of 3 tibial designs for patients undergoing TKA. Those results will be measured with disease-specific (Knee Society Scores), global (SF-36), and outcome measures. | 2 months, 1 year, 2 years, and 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Mark W. Pagnano, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States